CLINICAL TRIAL: NCT01960569
Title: Single Centre,Randomized,Phase IV Study to Assess the Topical r-Hirudin (Thrombexx)Efficacy in the Patients With Haematomas
Brief Title: Topical r-Hirudin ( Thrombexx ) Efficacy in Treatment of Haematomas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MinaPharm Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Minpharm07052012
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: r-Hirudin (Thrombexx) Efficacy in Treatment of Haematomas
Keywords: Thrombexx; Topical r-Hirudin; Efficacy; haematoma
MeSH Terms: conditions — Hematoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 : active product (Thrombexx) (Active Comparator): 100 patients will have the active product(Thrombexx), their visits on days 1,4,8 and 16 for target parameters assessment
  Interventions: Drug: active product ( Thrombexx) assigned to arm 1
- Arm 2 : Placebo (Placebo Comparator): 100 patients will have placebo , their visits on days 1,4,8 and 16 for target parameters assessment
  Interventions: Other: Placebo assigned to arm 2

INTERVENTIONS:
Drug: active product ( Thrombexx) assigned to arm 1 — Dispense 2-3 cm of cream or gel, 2-3 times per day and carry out a light massage until complete
  Other Names: Topical r-Hirudin
  Arms: Arm 1 : active product (Thrombexx)
Other: Placebo assigned to arm 2
  Arms: Arm 2 : Placebo

SUMMARY:
Single centre ,Phase IV , interventional, The study includes :

200 patients, 100 Patients will have Topical r-Hirudin (Thrombexx) and 100 patients will have placebo .

The patients will be randomized to the active product (arm 1) or to placebo (arm 2).

The study consists of 4 visits as the following :

* Visit 1 : on day 1 to check patient eligibility and also for randomization .
* Visit 2 : on day 4 to assess target parameters
* Visit 3 : on day 8 to assess target parameters
* Visit 4 : on day 16 to assess target parameters

DETAILED DESCRIPTION:
Single centre ,Phase IV , interventional, The study includes :

* 200 patients, 100 Patients will have Topical r-Hirudin (Thrombexx) and 100 patients will have placebo .

The patients will be randomized to the active product (arm 1) or to placebo (arm 2).

The study consists of 4 visits as the following :

* Visit 1 : on day 1 to check patient eligibility and also for randomization .
* Visit 2 : on day 4 to assess target parameters
* Visit 3 : on day 8 to assess target parameters
* Visit 4 : on day 16 to assess target parameters

  * Study objective :Assessment the Efficacy of Topical r-Hirudin in treatment of haematomas ,also in resolving of the associated oedema
  * Study duration : 6 months
  * Selection of trial subjects:

Inclusion Criteria :

1. Age of patients between 20 and 60 years old.
2. Patients with all types of haematomas.

Exclusion Criteria:

1. Presence of infected wound requiring hospitalization or surgical intervention.
2. History of allergy or hypersensitivity to any of the ingredients.
3. Patients with coagulation disorders like haemophilia.
4. Patients who are on anticoagulants like Warfarin and Acetylsalicylic acid .
5. Patients who are taking digestive enzymes like alfa chemotrypsin.

   * Target parameters :

1.Size of haematoma.( Measured by ruler) , The ruler will measure the longest 2 intersecting line.

2.Size of oedema : by measurement of oedema circumference

3.Pain (by Vas score).

4.Change in colour ( by colour grade scale ) .

ELIGIBILITY:
Inclusion Criteria:

* Age of patients between 20 and 60 years old.
* Patients with all types of haematoma.

Exclusion Criteria:

* Presence of infected wound requiring hospitalization or surgical intervention.
* History of allergy or hypersensitivity to any of the ingredients.
* Patients with coagulation disorders like haemophilia.
* Patients who are on anticoagulants like Warfarin and Acetylsalicylic acid .
* Patients who are taking digestive enzymes like alfa chemotrypsin.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Size of haematoma | 6 months
  Assessment the size of haematoma will be by ruler with unit centimeter(cm) , The ruler will measure the longest 2 intersecting line.
Size of oedema | 6 months
  Assessment the size of oedema will be by measurement the circumference in unit centimeter(cm).
Severity of Pain | 6 months
  Assessment of pain severity will be by Vas score
Change in Colour | 6 months
  Assessment of colour will be by colour grade scale , A=Bluish red , B=Blue ,C= Faint

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hafez, Professor, Principal Investigator — 6th October university; Ahmed Moneer, Dr, Study Chair — 6th october university
Locations (1):
- Prof. Mahmoud Hafez, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] El-Mowafi H, El Araby A, Kandil Y, Zaghloul A. Randomized, double-blind, placebo-controlled, interventional phase IV investigation to assess the efficacy and safety of r-hirudin gel (1120I.U) in patients with hematomas. Res Pract Thromb Haemost. 2017 Nov 6;2(1):139-146. doi: 10.1002/rth2.12049. eCollection 2018 Jan. PMID 30046714